CLINICAL TRIAL: NCT04663191
Title: Intraoperative Conversion During Video-assisted Thoracoscopy Resection for Lung Cancer Does Not Alter Survival
Acronym: ICVATR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: T38
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Video-assisted Thoracoscopic Surgery; Lung Cancer; Lobectomy; Survival; Surgery
Keywords: video-assisted thoracoscopic surgery; lung-cancer surgery; intraoperative conversion to open surgery; lobectomy; survival
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Full VATS
  Interventions: Procedure: anatomical resection
- VATS with conversion
  Interventions: Procedure: anatomical resection
- Thoracotomy upfront
  Interventions: Procedure: anatomical resection

INTERVENTIONS:
Procedure: anatomical resection — Anatomical resection with systematic lymph-node dissection

SUMMARY:
Anatomical resection with systematic lymph-node dissection is currently the standard of care for the treatment of early stage non-small cell lung cancer. The use of minimally invasive approaches has increased greatly over the last two decades [either video-assisted thoracoscopic surgery (VATS) or robotic-assisted thoracoscopic surgery (RATS)], as they provide the patient with better outcomes than open thoracotomy. Minimally invasive VATS lobectomy for a standard case is generally a straightforward procedure for a well-trained surgical team, although concomitant preoperative pathologies or intraoperative findings/adverse events may result in technical difficulties, leading to intraoperative conversion, commonly by thoracotomy.

The investigators aimed to assess long-term outcomes in a consecutive cohort of patients treated by anatomical pulmonary resection either using VATS, VATS requiring intraoperative conversion to thoracotomy, or upfront open thoracotomy for lung-cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients treated by anatomical lobar pulmonary resection (lobectomy, bilobectomy) or anatomical sublobar pulmonary resection (segmentectomy) for non-small cell lung cancer (NSCLC), either by VATS (eventually with intraoperative conversion) or upfront thoracotomy.

Exclusion Criteria:

* patients with non-anatomical pulmonary resection (wedge resection)
* patients with a histology other than NSCLC (benign or metastatic from another primitive cancer), stage IV NSCLC disease,
* patients with multiple primary NSCLC (synchronous or metachronous)
* patients with incomplete resection (R+)
* patient for whom a VATS approach was never considered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated by anatomical lobar pulmonary resection (lobectomy, bilobectomy) or anatomical sublobar pulmonary resection (segmentectomy) for non-small cell lung cancer (NSCLC), either by VATS (eventually with intraoperative conversion) or upfront thoracotomy.
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Overall survival during the follow-up period after surgery | from day of surgery up to 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No